CLINICAL TRIAL: NCT01067846
Title: The Clinical and Neural Response of Cocaine Addicts to Combination Treatment With a Cognitive Enhancer and Extinction-Based Psychotherapy
Brief Title: Cognitive Enhancement and Relapse Prevention in Cocaine Addiction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Arkansas (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 111989; R21DA025243 (NIH)
Record Dates: First submitted 2010-02-10; First posted 2010-02-12 (Estimated); Results first posted 2013-11-26 (Estimated); Last update posted 2013-11-26 (Estimated); Status verified 2013-10

CONDITIONS: Cocaine Addiction
Keywords: cocaine dependence; relapse prevention; computerized cognitive behavioral therapy (CBT); D-cycloserine (DCS)
MeSH Terms: conditions — Cocaine-Related Disorders | interventions — Cycloserine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- DCS and Cognitive Behavioral Therapy (Experimental): Subjects will receive 250 mg of Seromycin or D-cycloserine (DCS) prior to computerized cognitive behavioral therapy.
  Interventions: Drug: Seromycin (D-cycloserine, DCS); Behavioral: Computerized Cognitive Behavioral Therapy
- Placebo and Cognitive Behavioral Therapy (Placebo Comparator): Subjects will receive a 250 mg identical looking placebo pill prior to computerized cognitive behavioral therapy.
  Interventions: Drug: Placebo; Behavioral: Computerized Cognitive Behavioral Therapy

INTERVENTIONS:
Drug: Seromycin (D-cycloserine, DCS) — 250 mg DCS once weekly for 4 weeks prior to the initiation of a Computerized Cognitive Behavioral Therapy (CBT) session for drug relapse intervention.
  Other Names: D-cycloserine, DCS
  Arms: DCS and Cognitive Behavioral Therapy
Drug: Placebo — Placebo identical looking to the 250 mg DCS once weekly for 4 weeks prior to the initiation of a Computerized Cognitive Behavioral Therapy (CBT) session for drug relapse intervention.
  Arms: Placebo and Cognitive Behavioral Therapy
Behavioral: Computerized Cognitive Behavioral Therapy — All participants received Computerized Cognitive Behavioral Therapy sessions 3 times per week for 4 weeks as a drug relapse intervention.

SUMMARY:
For this project, the investigators are interested in exploring a new way to extend and maintain drug abstinence in people who are addicted to crack cocaine. This study will combine a medication called D-Cycloserine (DCS) and weekly cognitive behavioral therapy (CBT) to assess whether the combination will enhance people's ability to stay clean (drug free) for longer periods of time.

One of the greatest risks for drug relapse is drug craving. Oftentimes drug craving occurs when a person is confronted with stressors and reminders of past drug use behavior. DCS has been shown to enhance the learning of new information. By administering DCS prior to learning new techniques such as how to cope with drug craving and drug-use reminders, it is possible that patients can be more successful at living a drug free life for a longer period of time.

In addition to exploring this model behaviorally, the investigators will explore changes that may occur in the brain before and after the therapy/medication intervention. A technique called MRI (Magnetic Resonance Imaging) will be used to identify areas of the brain that are being activated during an attention task. Areas of neural activation will be assessed at study entry, end of therapy (4-week endpoint) and one month following completion of the treatment program.

DETAILED DESCRIPTION:
Primary Hypothesis:

Enhancing glutamatergic neurotransmission with DCS facilitates CBT-related relapse prevention by potentiating the behavioral and neural representation of the diminished drug motivation associated with cocaine cues.

Specific Aims:

1. Determine if the short-term oral administration of DCS relative to placebo prior to CBT sessions facilitates cocaine abstinence and functional recovery, and reduces cocaine craving in treatment-seeking cocaine addicts.
2. Determine if DCS administration relative to placebo facilitates CBT-related decreases in the behavioral and neural response to conditioned cocaine cues.

ELIGIBILITY:
Inclusion Criteria:

* Eligible subjects must be cocaine-dependent persons between 18 and 65 years

Exclusion Criteria:

* Any current Axis-I psychiatric diagnosis other than cocaine or alcohol dependence or nicotine use
* Any current or prior neurological disease, history of a major medical illness, or current use of psychotropic medications
* Positive history of loss of consciousness of greater than 10 min
* Significant current or prior cardiovascular disease (hypertension, arrhythmias) that is not medically stable
* History of hospitalization within the previous six months for a medical illness
* Deafness, blindness or other significant sensory impairment.
* Contraindications for D-cycloserine and magnetic resonance imaging.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 85 (Actual)
Dates: Start 2010-06; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinton Kilts, PhD, Principal Investigator — University of Arkansas
Locations (1):
- Psychiatric Research Institute (PRI) (Center for Addiction Research (CAR) and Brain Imaging Research Center (BIRC)) University of Arkansas for Medical Sciences, Little Rock, Arkansas, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment included outpatient and inpatient alcohol and drug abuse clinics, self-referrals, flyers in public places, and advertisements in newspapers. Recruitment started June 2010 and ended September 2011.
Pre-assignment Details: Enrolled participants could have been excluded due to other drug dependencies, loss of consciousness > 10 min, neurologic disorder, severe hepatic insufficiency, significant cardiovascular disease, current psychiatric disorder, current medical illness, sensory impairment, positive pregnancy test.
Groups:
- DCS and Cognitive Behavioral Therapy: Subjects will receive 250 mg of Seromycin or D-cycloserine (DCS) prior to computerized cognitive behavioral therapy.
  Seromycin (D-cycloserine, DCS) : 250 mg DCS once weekly for 4 weeks prior to the initiation of a Computerized Cognitive Behavioral Therapy (CBT) session for drug relapse intervention.
- Placebo and Cognitive Behavioral Therapy: Subjects will receive a 250 mg identical looking placebo pill prior to computerized cognitive behavioral therapy.
  Placebo : Placebo identical looking to the 250 mg DCS once weekly for 4 weeks prior to the initiation of a Computerized Cognitive Behavioral Therapy (CBT) session for drug relapse intervention.
Period: Overall Study
Arm/Group | DCS and Cognitive Behavioral Therapy | Placebo and Cognitive Behavioral Therapy
Started | 29 (Due to exclusion prior to group assignment, Study Enrollment will not equal Total # of Participants.) | 30 (Due to exclusion prior to group assignment, Study Enrollment will not equal Total # of Participants.)
Completed 3 Tx Sessions | 15 (Our final analysis includes these participants.) | 15 (Our final analysis includes these participants.)
Completed | 10 (Participants that completed all 4 weeks of treatment.) | 11 (Participants that completed all 4 weeks of treatment.)
Not Completed | 19 | 19
Not completed — Lost to Follow-up | 17 | 19
Not completed — Withdrawal by Subject | 1 | 0
Not completed — participation in other tx study | 1 | 0

BASELINE CHARACTERISTICS:
Population: These numbers include participants that were eligible after the initial intake assessment and were assigned to a group.
Groups:
- Total: Total of all reporting groups
Arm/Group | DCS and Cognitive Behavioral Therapy | Placebo and Cognitive Behavioral Therapy | Total
Number analyzed (Participants) | 29 | 30 | 59
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 29 | 30 | 59
  >=65 years | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 44 (6.67) | 45 (9.13) | 44 (7.97)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 4 | 11
  Male | 22 | 26 | 48
Region of Enrollment [Number; unit: participants]
  United States | 29 | 30 | 59

OUTCOME MEASURES:

1. Primary Outcome: Drug Abstinence During Treatment and at Follow up Visits
Description: Percentage of the overall number of drug abstinences of participants measured by urine drug testing
Time Frame: Participants provided urine samples for drug testing during treatment which occurred 3 times per week for 4 weeks, at the end of treatment, and at a 1 and 2 month follow up visit
Population: Total possible urine samples = 225 per arm. Not all participants stayed in treatment, therefore the total units analyzed will not match the total possible.
Measure: Number; unit: percentage of drug abstinences
Units Other Than Participants: Urine Samples
Arm/Group | DCS and Cognitive Behavioral Therapy | Placebo and Cognitive Behavioral Therapy
Number analyzed (Participants) | 15 | 15
Number analyzed (Urine Samples) | 181 | 188
percentage of drug abstinences | 12 | 25

2. Primary Outcome: Treatment Retention - Number of Visits During Treatment
Description: Number of treatment visits attended prior to discontinuation of treatment
Time Frame: Treatment sessions included 3 visits per week for 4 weeks
Population: Total possible sessions attended = 180 per arm. Some participants did not complete all sessions, therefore the units analyzed will not match the total possible.
Measure: Mean (Standard Deviation); unit: visits
Units Other Than Participants: Sessions Attended
Arm/Group | DCS and Cognitive Behavioral Therapy | Placebo and Cognitive Behavioral Therapy
Number analyzed (Participants) | 15 | 15
Number analyzed (Sessions Attended) | 149 | 150
visits | 10 (3) | 10 (3)

ADVERSE EVENTS:
Time Frame: 1 year, 7 months
Arm/Group | DCS and Cognitive Behavioral Therapy | Placebo and Cognitive Behavioral Therapy
Serious Adverse Events (participants affected / at risk) | 0/29 | 0/30
Other Adverse Events (participants affected / at risk) | 3/29 | 2/30
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | DCS and Cognitive Behavioral Therapy (N=29) | Placebo and Cognitive Behavioral Therapy (N=30)
cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) — Participant reported infrequent coughing. Physician determined it was not study related.
headache (Nervous system disorders) | 1 (1) | 0 (0) — Participant reported mild headaches. Physician determined it was not study related.
nausea (General disorders) | 1 (1) | 0 (0) — Participant reported a nauseas feeling. Physician determined it was not study related.
sensation on skin (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2) — Participant reported a crawling sensation on skin. Physician determined it was not study related.
rash on skin (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2) — Participant reported a rash on skin. Physician determined it was not study related.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No